CLINICAL TRIAL: NCT07180355
Title: A Phase 1b First-in-Human, Open-Label, Dose-Finding Trial to Evaluate the Safety and Tolerability of SGT-212 Delivered Via Dual Intradentate Nucleus (IDN) and Intravenous (IV) Administration to Participants With Friedreich's Ataxia (FA)
Brief Title: A Study of SGT-212 Gene Therapy in Friedreich's Ataxia
Acronym: FALCON
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Solid Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGT-212-101
Record Dates: First submitted 2025-08-22; First posted 2025-09-18 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Friedreich's Ataxia (FA)
Keywords: SGT-212; Gene Therapy; Frataxin; Repeat Expansion; Neuromuscular; Cardiac; Ataxia; Movement Disorder; Rare disease; AAV; AAVhu68
MeSH Terms: conditions — Friedreich Ataxia; Ataxia; Movement Disorders; Rare Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Non-Ambulatory) (Experimental): Non-ambulatory participants will receive bilateral intradentate infusion (IDN) followed by systemic intravenous (IV) infusion.
  Interventions: Drug: SGT-212
- Cohort 2 (Ambulatory) (Experimental): Ambulatory participants will receive bilateral IDN infusion followed by systemic IV infusion.
  Interventions: Drug: SGT-212
- Cohort 3 (Ambulatory and Non-Ambulatory) (Experimental): Participants will receive bilateral IDN followed by systemic IV infusion.
  Interventions: Drug: SGT-212

INTERVENTIONS:
Drug: SGT-212 — Adeno-associated virus serotype AAVhu68 containing a codon-optimized complementary DNA (cDNA)

SUMMARY:
This is a phase 1b, first in-human, open-label, dose-finding study investigating the safety and tolerability of SGT-212 in participants with Friedreich's ataxia (FA). It will be delivered via dual intradentate nucleus (IDN) and intravenous (IV) administration to participants with FA.

All participants will receive SGT-212 and will be enrolled in the study for approximately 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Has history of FA symptom onset ≤25 years of age
* Has a clinical and genetic diagnosis of FA
* Has a staging score of ≥1 but <6 on the Friedreich's Ataxia Rating Scale (FARS) Functional Disability Staging Score
* Is willing to agree to the following rules for use of omaveloxolone (Skyclarys):

  1. For a candidate who is currently taking omaveloxolone, has been on a stable dose for 12 weeks, expects to continue taking omaveloxolone at that dose throughout the study, and is willing to stop taking omaveloxolone at the direction of the Investigator or Sponsor's Medical Monitor if evidence of transaminitis or synthetic liver dysfunction is detected during the study
  2. For a candidate who is not actively taking omaveloxolone, at least 12 weeks have passed since the last dose and the candidate agrees not to resume omaveloxolone during the 18-month period after SGT-212 infusion NOTE: The use of any other approved or investigational medicinal product for the treatment of FA should be discussed with the study team.

Exclusion Criteria:

* Antibodies against adeno-associated virus serotype 9 (AAV9)
* Has a modified FARS (mFARS) score <20
* Has a body weight ≤25 kilogram (kg) or has body mass index (BMI) ≥33 kg/m^2
* Has a contraindication to endomyocardial biopsy (EMB) or cardiac catheterization
* Is unable to undergo cardiac and brain MRI with contrast, including hypersensitivity to gadolinium contrast agent, presence of a non-MRI-compatible cardiac pacemaker, presence of a non-MRI-compatible implantable cardiac defibrillator, or physical condition (e.g., contractures)
* Has uncontrolled diabetes as defined by a hemoglobin (Hb) A1c >9%
* Has participated in recent interventional clinical studies or received any investigational therapy administered within 3 months or 5 half-lives (whichever is longer) prior to Screening
* Has received gene therapy at any time
* Has contraindications to receiving corticosteroids
* Has any contraindication to the surgical procedures involved with IDN infusion of SGT-212
* Has any known cardiac disease not related to FA including known obstructive coronary artery disease (CAD)
* Other Inclusion/Exclusion criteria to be applied as per protocol.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2028-03-21 (Estimated); Study Completion 2032-02-29 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Treatment Emergent Adverse Events (TEAEs) | Month 12

SECONDARY OUTCOMES:
Incidence and Severity of TEAEs | Months 18 and 60
Incidence and Severity of Treatment-emergent Serious adverse events (SAEs) | Months 18 and 60
Number of Treatment-emergent deaths | Months 18 and 60
Change from Baseline in Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline, Months 18 and 60
Number of Participants with Change from Baseline in Significant Abnormalities in Laboratory Tests | Baseline, Months 18 and 60
Number of Participants with Change from Baseline in Significant Abnormalities in Vital Signs | Baseline, Months 18 and 60
Number of Participants with Change from Baseline in Significant Abnormalities in Physical Examination Findings | Baseline, Months 18 and 60
Number of Participants with Change from Baseline in Innate and Adaptive Immune Responses | Baseline, Months 18 and 60
Change from Baseline in Blood Biomarkers Including Inflammatory Markers | Baseline, Month 12

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The Ohio State University, Columbus, Ohio
  - The Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No